CLINICAL TRIAL: NCT01800565
Title: Urinary LH in the Diagnosis of Precocious Puberty
Brief Title: First-Voided Urinary LH vs. GnRH-stimulation in Differentiating Slowly- From Rapidly Progressive-Precocious Puberty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amnon Zung (Other)
Responsible Party: Sponsor-Investigator, Amnon Zung, MD, Kaplan Medical Center
Organization: Kaplan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ULH
Record Dates: First submitted 2013-02-21; First posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Precocious Puberty, Gonadotropin-dependent
Keywords: precocious puberty; urinary LH; GnRH stimulation test; gonadotropins
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pubertal progression (Other): A collection of first voided urine sample for the measurement of LH.
  Interventions: Other: Measurement of LH in first-voided urine; Other: collection of first-voided urine sample for LH level

INTERVENTIONS:
Other: Measurement of LH in first-voided urine — participants in this study will be studied by the standard GnRH stimulation test. In addition, they will provide first voided urine sample (the experimental part)for the measurement of LH.
Other: collection of first-voided urine sample for LH level — participants in this study will be studied by the standard GnRH stimulation test. In addition, they will provide first voided urine sample (the experimental part)for the measurement of LH.

SUMMARY:
Precocious puberty (PP) in girls is classically defined by the onset of secondary sexual characteristics before eight years of age, but subsequent pubertal maturation can be quite varied. In many girls, PP takes a rapid course of progression (rapidly progressive precocious puberty; RP-PP) with an early menarche and fusion of the epiphyseal growth plates, leading eventually to a reduced final height if not treated. In a subset of girls with PP however, the growth rate slows to normal for age, skeletal maturation progresses in accordance with chronological age and there is little to no risk of impairment of final height (slowly progressive precocious puberty; SP-PP). Other conditions of non-progressive PP include premature breast budding and unsustained PP that is characterized by a spontaneous regression of sexual precocity. Due to their benign course, slowly progressive (SP) PP and other non-progressive forms of PP do not warrant therapy with GnRH agonists. Differentiating these forms from RP-PP is therefore essential to prevent unnecessary intervention in a population that accounts for at least 50% of girls with PP. A distinction between these forms of PP may be difficult on clinical grounds however, since all these patients may present initially as isolated breast development.

The gold standard for the diagnosis of true (central) PP is the measurement of gonadotropins following GnRH stimulation test. There is however an overlap between prepubertal and early pubertal values and between girls with premature breast budding and progressive PP. It was suggested therefore that progressive pubertal development and growth acceleration should be documented over a 3- to 6-months period before GnRHa therapy in initiated.

More than a decade ago several studies demonstrated that urinary gonadotropins are age related and significantly increased during puberty. It has been suggested that urinary gonadotropins measurements can be used for differential diagnosis of pubertal disorders. This is based on the assumption that gradual elevation of nocturnal LH secretion prior to and at the onset of puberty can be reflected by first-voided urinary LH (ULH). In this prospective study, the investigators aimed to evaluate the value of first-voided ULH measurements in predicting pubertal course and differentiating SP-PP from RP-PP, by comparison to GnRH-stimulated gonadotropins.

DETAILED DESCRIPTION:
Precocious puberty (PP) in girls is classically defined by the onset of secondary sexual characteristics before eight years of age, but subsequent pubertal maturation can be quite varied. In many girls, PP takes a rapid course of progression (rapidly progressive precocious puberty; RP-PP) with an early menarche and fusion of the epiphyseal growth plates, leading eventually to a reduced final height if not treated. In a subset of girls with PP however, the growth rate slows to normal for age, skeletal maturation progresses in accordance with chronological age and there is little to no risk of impairment of final height (slowly progressive precocious puberty; SP-PP). Other conditions of non-progressive PP include premature thelarche and unsustained PP that is characterized by a regression of sexual precocity. Due to their benign course, slowly progressive (SP) PP and other non-progressive forms of PP do not warrant therapy with GnRH agonists. Differentiating these forms from RP-PP is therefore essential to prevent unnecessary intervention in a population that accounts for at least 50% of girls with PP. A distinction between these forms of PP may be difficult on clinical grounds however, since all these patients may present initially as isolated breast development.

The gold standard for the diagnosis of true (central) PP is the measurement of gonadotropins following GnRH stimulation test , where peak LH and peak LH/FSH ratio are the most valuable diagnostic parameters. There is however an overlap between prepubertal and early pubertal values and between girls with premature thelarche and progressive PP. It was suggested therefore that progressive pubertal development and growth acceleration should be documented over a 3- to 6-months period before GnRHa therapy in initiated.

More than a decade ago, along with the development of high-sensitive immunoassay for gonadotropins that replaced the RIA, Demir and colleagues have shown that urinary gonadotropins are age related and significantly increased during puberty. It has been suggested by others that urinary gonadotropins measurements can be used for differential diagnosis of pubertal disorders. This is based on the assumption that gradual elevation of nocturnal LH secretion prior to and at the onset of puberty can be reflected by first-voided urinary LH (ULH). In this prospective study, the investigators aimed to evaluate the value of first-voided ULH measurements in predicting pubertal course and differentiating SP-PP from RP-PP, by comparison to GnRH-stimulated gonadotropins.

ELIGIBILITY:
Inclusion Criteria:

* Onset of puberty after 3 years of age in boys and girls
* Onset of puberty before 8 years in girls and 9 years in boys

Exclusion Criteria:

* Non-central precocious puberty
* Congenital adrenal hyperplasia
* Enuresis nocturne

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Estimated)
Dates: Start 2006-06; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Identification of first-voided urinary LH cutoff for the detection of pubertal advancement by comparison with GnRH stimulated gonadotropins | 2 years

SECONDARY OUTCOMES:
Levels first-voided urinary LH measurements in monitoring gonadotropin suppression during GnRHa therapy | 2 years

OTHER OUTCOMES:
Identification of first-voided urinary LH cutoff for differentiating pseudothelarche from true breast budding, compared with GnRH stimulated gonadotropins | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Amnon Zung, MD, Principal Investigator — Pediatirc Endocrinology Unit, Kaplan Medical Center, affiliated with the Hebrew University of Jerusalem, Israel
Locations (1):
- Peditaric Endocrinology Unit, Kaplan Medical Center, Rehovot, Israel